CLINICAL TRIAL: NCT03327155
Title: Western Australian Pre-exposure Prophylaxis for HIV Implementation Trial
Acronym: PrEPIT-WA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Government of Western Australia, Department of Health (Unknown); Western Australia AIDS Council (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HEPP1701
Record Dates: First submitted 2017-09-08; First posted 2017-10-31 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: HIV Prevention
Keywords: HIV prevention; PrEP
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: The study is proposed as implementation research to mimic the conditions that will occur when PrEP is rolled out at the population level. However, as the version of TDF/FTC used in this study, manufactured by Mylan, is not approved for use as PrEP in Australia, the study is conducted under the Clinical Trial Notification (CTN) scheme and within the CTN framework. After collection of consent and enrolment information, all follow-up information will be collected through electronic data capture to allow accurate and timely analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TDF/FTC (300mg/200mg) once daily (Experimental): Tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) (300mg/200mg) on tablet once daily with food.
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC)

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) — One tablet, containing 300mg of TDF and 200mg of FTC once daily with food.
  Other Names: TDF/FTC

SUMMARY:
Despite all prevention efforts, many people in Australia continue to be infected with HIV. The Seventh National HIV Strategy 2014-2017 in Australia aims to work towards the elimination of HIV transmission by the year 2020. This project will evaluate a new additional way to lower people's chances of getting HIV. It will provide pre-exposure prophylaxis (PrEP) to people who are at high risk for HIV and evaluate what impact this new prevention approach will have on HIV in WA at the community level.

The drug used in PREPIT-WA is called generic TDF/FTC (made by Mylan Laboratories Ltd.). The generic TDF/FTC is a single tablet made up of two HIV medications: tenofovir disoproxil fumarate and emtricitabine (a combination known as TDF/FTC). TDF and FTC have been widely used for many years to treat HIV. When used with other medicines in people who already have HIV, TDF/FTC reduces the amount of HIV virus in the blood. TDF/FTC does not cure HIV or AIDS, and it is not an HIV vaccine.

As a treatment for people who already have HIV, TDF/FTC is approved for use in most of the world, including Australia. As a medicine for PrEP, to lower chances of HIV in those who are not infected, TDF/FTC has been approved in the US, and Truvada® (which contains TDF/FTC made by Gilead Sciences Inc.) was approved for PrEP in Australia in May 2016. At the start of the project, the generic TDF/FTC is not approved in Australia for the use as PrEP but it may become registered for use and more freely available in Australia in the future.

DETAILED DESCRIPTION:
The Australian seventh National HIV strategy (2014-2017) aims to reduce the incidence of HIV and to work towards the virtual elimination of HIV transmission in Australia by 2020. This extraordinary goal relies on two anti-retroviral therapy (ARV)-related interventions, in addition to traditional behavioural prevention. The first of these interventions, HIV treatment as prevention targeted at HIV positive people, has been ramped up over the last few years, and is approaching maximal levels of population impact. Despite this, new HIV diagnoses in Australia have been approximately constant over the last four years. Critical to the new strategy's success is the population-based, targeted roll-out of HIV PrEP. PrEP involves taking one pill daily of co-formulated tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC). TDF/FTC has been extensively used in millions of people with HIV for more than 15 years.

This large-scale study aims for the rapid roll-out of TDF/FTC to individuals at high risk of HIV, who will comprise mostly gay and bisexual men (GBM) but will also include small numbers of heterosexuals, people who inject drugs, and transgender men and women. The drug will be used according to existing Australasian Society for HIV, Viral Hepatitis and Sexual Health (ASHM) HIV PrEP Clinical Guidelines.

By rapidly rolling out this new intervention as rapidly as feasible, and following participants for up to two years on treatments, we expect a reduction in new HIV diagnoses in WA due to decreased infection in the on-treatment cohort, and to the interruption of chains of transmission to others not receiving PrEP. The rapid and large-scale roll-out of PrEP is a critical component of working towards the virtual elimination of HIV transmission by 2020.

ELIGIBILITY:
Inclusion Criteria:

1. HIV negative at enrolment, with a negative HIV test result conducted at the enrolment clinic within seven days of initiating PrEP
2. At high and ongoing risk for acquiring HIV infection [as defined by Behavioural Eligibility criteria in the Australasian Society for HIV, Viral Hepatitis and Sexual Health Medicine (ASHM) HIV PrEP Clinical Guidelines]
3. Aged 18 years or over
4. Live in WA or visit WA enough to attend clinics for follow-up assessments
5. Willing and able to provide informed consent
6. Medicare ineligible individuals may be enrolled if the clinical service is able to cover the costs of monitoring of the patient

Exclusion Criteria:

1. HIV-1 infected or has symptoms consistent with acute viral infection (If HIV positive status is not confirmed by testing, delay starting PrEP for at least one month and reconfirm negative HIV-1 status)
2. Having an estimated creatinine clearance (glomerular filtration rate [eGFR]) <60ml/min
3. Having or developing clinical symptoms suggestive of lactic acidosis or pronounced hepatotoxicity (including nausea, vomiting, unusual or unexpected stomach discomfort, and weakness)
4. Concurrently taking a nephrotoxic agent (e.g., high-dose non-steroidal anti-inflammatory drugs / NSAIDs)
5. Allergic to TDF and/or FTC (based on self-report or recorded)
6. Concurrently taking prescribed products containing FTC or TDF including ATRIPLA®, COMPLERA®, EMTRIVA, STRIBILD®, VIREAD, TAF (tenofovir alafenamide), GENVOYA, DESCOVY; other drugs containing lamivudine; HEPSERA
7. Factors or conditions that may compromise a participant's access to health services for follow-up (incarceration or planned relocation and potential absence from Western Australia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of HIV infection per 100 person years among study participants | 24 weeks after the last participant completed their last follow-up visit (Month 18 visit)
  Statistical analyses of risk of HIV seroconversion among individuals who were prescribed PrEP (as part of the study) will focus on estimating the risk of seroconversion per 100 person years after TDF/FTC prescription and the effect modifying role of non-adherence to the prescribed medication schedule.
Number of HIV diagnoses among gay and bisexual men notified to Western Australian Department of Health | number of HIV diagnoses in the 12 month period prior to the date of first recruitment will be compared to the annual number of HIV diagnoses in the 12 month period after the study is fully recruited
  Number of diagnoses will be measured using routinely reported data from the Western Australia registry of HIV diagnoses

SECONDARY OUTCOMES:
Trends in test positivity of Sexually Transmitted Infections (STIs, gonorrhoea, chlamydia and infectious syphilis) among study participants | 24 weeks after the last participant completed their last follow-up visit (Month 18 visit)
  To calculate trends in test positivity of STI (gonorrhoea, chlamydia and infectious syphilis) among study participants, and describe changes over time
Number of enrollment to the study by clinic type | up to 6 months
  To measure in the four study sites

CONTACTS AND LOCATIONS:
Overall Officials: David Cooper, MD, Study Chair — The Kirby Institute, UNSW Sydney; Andrew Grulich, MBBS, MSc (Epid), PhD, Study Chair — The Kirby Institute, UNSW Sydney
Locations (4):
- Australia (4):
  - South Terrace Sexual Health Clinic, Fremantle, Western Australia
  - GP on Beaufort, Mount Lawley, Western Australia
  - Royal Perth Hospital Sexual Health Clinic, Perth, Western Australia
  - M Clinic, Perth, Western Australia